# PEERS Plus - mHealth Enhanced Peer Support to Reduce Depression Among Low-income and Ethnic Minority Older Adults

Study Protocol

NCT05611996

May 1<sup>st</sup>, 2025

#### Study:

Feasibility pilot study with approximately 32 participants Preliminary analysis of primary (PHQ-9) and secondary outcomes.

### **Statistical Analysis**

Baseline characteristics, working alliance scores, and clinical and social outcomes were summarized. The Shapiro-Wilk test was applied to check the normality of each outcome measure. Paired-sample t-tests and Wilcoxon signed-rank test were conducted to assess the differences in outcome measures between baseline and post-study, as well as baseline and three-month follow-up scores, to determine statistical significance. For all analyses, a significance level of alpha = 0.05 was used for two-sided tests unless otherwise specified.

To assess the change in the primary outcome, depressive symptoms over time within the intervention group, a multilevel linear regression model was employed. This model included fixed effects for time points (e.g., baseline, post-intervention, and follow-ups) and covariates such as baseline loneliness, self-efficacy, working alliance scores, and demographic variables that might influence the intervention effects. Random intercepts and slopes were included to account for the repeated measures within participants, allowing for individual variability in both baseline levels and the trajectories of depressive symptoms over time. Additionally, random effects were specified at the peer coach level to account for the nested structure of the data, where participants were grouped by peer coaches. These analyses and data visualizations were conducted using R Statistical Software (v4.2.1; R Core Team 2022).

# PHQ\_9

| 1110_0 | | | | | | Effect | |
|---|---|---|---|---|---|---|---|
| | | | 0 | | | Size(standardiz | |
| | | | Std. | | p- | | Marginal |
| Model | Timepoint | Estimate | Error | 95% CI | Value | coefficients) | R^2 |
| | Baseline vs | | | | | | |
| Model 1: Basic | Poststudy | -1.93 | 0.79 | (-3.513, -0.344) | 0.018 | -0.36 | 0.049 |
| | Baseline vs 3- | | | | | | |
| | mons follow- | | | | | | |
| | up | -2.88 | 0.83 | (-4.557, -1.209) | 0.001 | -0.54 | |
| Model 2: | | | | | | | |
| Adjusted for | | | | | | | |
| demographics | Baseline vs | | | | | | |
| # | Poststudy | -1.93 | 0.79 | (-3.509, -0.348) | 0.018 | -0.36 | 0.159 |
| | Baseline vs 3- | | | | | | |
| | mons follow- | | | | | | |
| | up | -2.81 | 0.83 | (-4.488, -1.137) | 0.001 | -0.53 | |
| Model 3: Full | Baseline vs | | | | | | |
| Model ## | Poststudy | -1.78 | 0.77 | (-3.336, -0.230) | 0.025 | -0.33 | 0.276 |
| | Baseline vs 3- | | | | | | |
| | mons follow- | | | | | | |
| | ир | -2.42 | 0.81 | (-4.057, -0.784) | 0.005 | -0.45 | |

<sup>#</sup> Model 2 adjusted for age, gender, education, marital status, race, and employment status.

## Self-Efficacy

| oet Emedey | | | | | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | Effect | |
| | | | Std. | | p- | Size(standardized | |
| Model | Timepoint | Estimate | Error | 95% CI | Value | coefficients) | Marginal R^2 |
| Model 1: | Baseline vs | | | | | | |
| Basic | Poststudy | 2.030 | 0.824 | (0.375, 3.686) | 0.017 | 0.40 | 0.051 |
| | Baseline vs | | | | | | |
| | 3-mons | | | | | | |
| | follow-up | 2.773 | 0.870 | (1.024, 4.521) | 0.003 | 0.55 | |
| Model 2: | | | | | | | |
| Adjusted for | | | | | | | |
| demographics | Baseline vs | | | | | | |
| # | Poststudy | 2.018 | 0.823 | (0.363, 3.673) | 0.018 | 0.40 | 0.383 |

<sup>##</sup> Model 3 adjusted for demographic variables and loneliness.

| | Baseline vs | | | | | | |
|---|---|---|---|---|---|---|---|
| | 3-mons<br>follow-up | 2 773 | 0 872 | (1.021, 4.525) | 0.003 | 0.55 | |
| | Baseline vs | | 0.072 | (1.021, 4.020) | 0.000 | 0.00 | |
| Model ## | Poststudy | 1.823 | 0.760 | (0.295, 3.351) | 0.020 | 0.48 | 0.566 |
| | Baseline vs | | | | | | |
| | 3-mons | | | | | | |
| | follow-up | 2.318 | 0.799 | (0.711, 3.926) | 0.006 | 0.55 | |

<sup>#</sup> Model 2 adjusted for age, gender, education, marital status, race, and employment status.

# **Emotional Well-being**

| Linotionat wet | 1 | 1 | 1 | | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | Effect | |
| | | | Std. | | p- | Size(standardized | |
| Model | Timepoint | Estimate | Error | 95% CI | Value | coefficients) | Marginal R^2 |
| Model 1: | Baseline vs | | | | | | |
| Basic | Poststudy | 6.571 | 2.668 | (1.208, 11.935) | 0.017 | 0.32 | 0.057 |
| | Baseline vs | | | | | | |
| | 3-mons | | | | | | |
| | follow-up | 12.566 | 2.869 | (6.801, 18.330) | 0.000 | 0.61 | |
| Model 2: | | | | | | | |
| Adjusted for | | | | | | | |
| demographics | Baseline vs | | | | | | |
| # | Poststudy | 6.571 | 2.663 | (1.220, 11.923) | 0.017 | 0.32 | 0.215 |
| | Baseline vs | | | | | | |
| | 3-mons | | | | | | |
| | follow-up | 12.293 | 2.870 | (6.526, 18.060) | 0.000 | 0.60 | |
| Model 3: Full | Baseline vs | | | | | | |
| Model ## | Poststudy | 5.375 | 2.593 | (0.159, 10.591) | 0.044 | 0.26 | 0.289 |
| | Baseline vs | | | | | | |
| | 3-mons | | | | | | |
| | follow-up | 11.119 | 2.784 | (5.519, 16.720) | 0.000 | 0.54 | |

<sup>#</sup> Model 2 adjusted for age, gender, education, marital status, race, and employment status.

## **Social Function**

| Model | Timepoint | | Std.<br>Error | | p- | Effect<br>Size(standardized<br>coefficients) | Marginal R^2 |
|---|---|---|---|---|---|---|---|
| Model 1: | Baseline vs | | | (- | | | |
| Basic | Poststudy | 5.804 | 4.656 | 3.557, 15.164) | 0.219 | 0.20 | 0.068 |

<sup>##</sup> Model 3 adjusted for demographic variables and loneliness.

<sup>##</sup> Model 3 adjusted for demographic variables and loneliness.

| | Baseline vs | | | | | | |
|---|---|---|---|---|---|---|---|
| | 3-mons | | | | | | |
| | follow-up | 18.775 | 4.994 | (8.740, 28.809) | 0.001 | 0.65 | |
| Model 2: | | | | | | | |
| Adjusted for | | | | | | | |
| demographics | Baseline vs | | | (- | | | |
| # | Poststudy | 5.804 | 4.648 | 3.539, 15.146) | 0.218 | 0.20 | 0.304 |
| | Baseline vs | | | | | | |
| | 3-mons | | | | | | |
| | follow-up | 18.385 | 5.004 | (8.329, 28.441) | 0.001 | 0.64 | |
| Model 3: Full | Baseline vs | | | (- | | | |
| Model ## | Poststudy | 5.926 | 4.612 | 3.350, 15.202) | 0.205 | 0.21 | 0.385 |
| | Baseline vs | | | | | | |
| | 3-mons | | | | | | |
| | follow-up | 16.447 | 4.944 | (6.504, 26.390) | 0.002 | 0.57 | |

<sup>#</sup> Model 2 adjusted for age, gender, education, marital status, race, and employment status.

<sup>##</sup> Model 3 adjusted for demographic variables and loneliness.